CLINICAL TRIAL: NCT06794242
Title: Investigating the Link Between Body Representation and Neuropathic Pain in Patients with Spinal Cord Injury
Brief Title: Body Representation and Neuropathic Pain in Spinal Cord Injury
Acronym: REPTAILLE
Status: Not yet recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: Centre de Recherche de Neurosciences de Lyon (Unknown)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0460
Record Dates: First submitted 2025-01-21; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Spinal Cord Injury
Keywords: Neuropathic pain; Spinal cord injury; Body representation; Virtual reality; Quality of life
MeSH Terms: conditions — Spinal Cord Injuries; Neuralgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients: Spinal cord injury subjects
  Interventions: Other: Body representation
- Controle: Healthy Subjects
  Interventions: Other: Body representation

INTERVENTIONS:
Other: Body representation — All the participants (controls and patients) in the study will follow the same experimental procedure, which consists of a single virtual reality session involving the estimation of leg length and an object.

SUMMARY:
Chronic pain is one of the main complications of spinal cord injury, has a very negative impact on quality of life, and persists over time despite the use of analgesic treatments. Several types of pain are possible in patients with spinal cord injury, and neuropathic pain (pain caused by damage to the spinal cord, in this case) is one of the most difficult to treat, even with medication. Following an injury to the spinal cord, it is possible for the representation of the body to change as a result of sensorimotor deficits, prolonged changes in body posture and altered mobility. At present, the causes of chronic pain after spinal cord injury remain poorly understood and debated, but one hypothesis suggests that changes in body representation may play a key role in the development or worsening of neuropathic pain. To test this hypothesis, we will assess the perception of spinal cord injured patients (and a group of controls) of the size of their legs using a virtual reality device. This measurement will enable us to examine whether under- or over-estimation of leg length correlates with the presence of neuropathic pain in patients. Chronic pain in people with spinal cord injury is associated with an increased risk of stress, depression and anxiety, and understanding and treating neuropathic pain in people with spinal cord injury is a major issue in their management.

ELIGIBILITY:
Inclusion Criteria :

Patients group:

* Men and women between the ages of 18 and 65;
* Have normal or corrected eyesight;
* Have a spinal cord lesion resulting in total or partial loss of tactile and proprioceptive sensitivity and motor skills in the lower limbs.
* have given their free and informed consent in writing, after having been informed orally and in writing of the study's progress.

Control group:

* Men and women between 18 and 65 years of age
* Have normal or corrected eyesight
* Have given their free and informed written consent after having been informed orally and in writing of the course of the study.

Exclusion Criteria :

Patients Group:

* People with a diagnosis of Eating Disorder
* People with a diagnosis of a psychiatric disorder that can modify body representations
* People who suffer from physiological discomfort when using gaming headsets or virtual reality
* People under psychiatric care
* Illiterate people
* Pregnant women, women in labour or breastfeeding mothers
* Persons deprived of their liberty by judicial or administrative decision
* Adults under legal protection (guardianship, curatorship)
* Persons not affiliated to a social security scheme or beneficiaries of a similar scheme

Control group:

* People with an eating disorder diagnosis
* People diagnosed with psychiatric disorders that can modify body representations
* People who suffer from physiological discomfort when using gaming headsets or virtual reality
* People under psychiatric care
* Illiterate people
* People with functional neurological motor disorders and/or partial or complete deficits and/or abnormal movements
* People with sensitivity problems in the lower limbs
* Pregnant women, women in labour or breastfeeding mothers
* Persons deprived of their liberty by judicial or administrative decision
* Persons admitted to a health or social establishment for purposes other than research
* Adults under legal protection (guardianship, curatorship)
* Persons not affiliated to a social security scheme or beneficiaries of a similar scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Spinal cord injury and volontary subjects
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Différences in leg length estimation between controls and patients in the length representation test. | From baseline up to a maximum of 2 weeks
  We will measure the difference between the representation of the length of the lower limbs of controls and spinal cord injured patients. This difference will be assessed using the Point of Subjective Equality (defined as the size of the avatar's legs perceived by the participant as corresponding to the length of their legs) with a two-sample Mann Whitney test (two-tailed) (controls and patients)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Pierre Wertheimer Neurological Hospital, Bron, France
  - Henry Gabrielle Hospital, Saint-Genis-Laval, France

IPD SHARING:
Plan to Share IPD: Undecided